CLINICAL TRIAL: NCT03100357
Title: Changes in Esophageal Motility and Swallowing Symptoms After Thyroid Surgery - a Prospective Cohort Study
Brief Title: Changes in Esophageal Motility and Swallowing Symptoms After Thyroid Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Jesper Roed Sorensen, MD PhD fellow, University of Southern Denmark
Other Study IDs: SOLOIST4
Record Dates: First submitted 2017-03-14; First posted 2017-04-04 (Actual); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Esophageal Motility Disorders
MeSH Terms: conditions — Esophageal Motility Disorders | interventions — Thyroidectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Thyroidectomy — Thyroid surgery for benign nodular goiter

SUMMARY:
The pronounced effect of goiter on the esophagus needs further exploration, as the mechanisms by which goiter leads to swallowing difficulties are unknown. By investigating esophageal motility using high resolution esophageal manometry before and after thyroidectomy we seek to examine the impact of the goiter mass on the esophagus and swallowing with six months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic benign nodular goiter referred for thyroidectomy

Exclusion Criteria:

* Previous surgery to the neck;
* Suspicion of thyroid cancer
* Age below 20 years or above 80 years
* Neuromuscular disease.

Ages: 20 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with benign nodular goiter
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Motility disturbances | Before and six months following thyroidectomy
  Change in number of failed swallowings from baseline

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sorensen JR, Markoew S, Dossing H, Hegedus L, Bonnema SJ, Godballe C. Changes in Swallowing Symptoms and Esophageal Motility After Thyroid Surgery: A Prospective Cohort Study. World J Surg. 2018 Apr;42(4):998-1004. doi: 10.1007/s00268-017-4247-5. PMID 29043407